CLINICAL TRIAL: NCT05530005
Title: Comparison of the Traditional Physiotherapy Protocol With Monitoring Individually Prescribed Exercises in Impingement Syndrome of the Shoulder Joint
Brief Title: Traditional Physiotherapy Protocol vs Prescribed Exercises in Impingement Syndrome of the Shoulder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Klinika Ruchu (Other)
Collaborators: Józef Piłsudski University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SKE01-11/2022
Record Dates: First submitted 2022-08-04; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: Subacromial Impingement Syndrome
Keywords: subacromial bursa; impingement syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hands on (Active Comparator): Patients with shoulder impingement syndrome. Age 18-50 years. Shoulder pain lasting from 3 months to 1 year, No surgery and injection intervention in the shoulder joint and surrounding area in the history of the disease. - Ailments in scales I and II according to Neer.
  Interventions: Other: Manual Therapy
- Hands off (No Intervention): Patients with shoulder impingement syndrome. Age 18-50 years. Shoulder pain lasting from 3 months to 1 year, No surgery and injection intervention in the shoulder joint and surrounding area in the history of the disease. - Ailments in scales I and II according to Neer.

INTERVENTIONS:
Other: Manual Therapy — Manual Therapy according to Kaltenborn Evjenth method. Exercises with PT resistance, massage.
  Arms: Hands on

SUMMARY:
Pain and limitation of shoulder mobility resulting from sub-shoulder syndrome called sub acromion impingement syndrome (SIS) are a big social problem in highly developed countries. This work aims to compare the method of treating SIS ailments taking into account the monitored exercises on their own- hands off, to the traditional method of individual physiotherapy considering manual therapy, TENS and local cryotherapy- hands on. The study will qualify people aged 18-50 years without previous injections, surgical procedures and physiotherapy within the shoulder joint. The initial examination of the participants will include: ultrasound examination, Neer test, functional mobility test according to FMS, clinical examination: palpation of the joint area, cross body adduction test, radial artery pulse test, numerical pain scale 0-10, DASH questionnaire. After the initial checkups, 60 people will be qualified for the proper examination. Selected participants will be divided into two groups of 30 people, each group consisting of 15 women and 15 men. The first group will undergo self-therapy for 3-5 months. The subjects will exercise independently for about 1.5 hours a day, three times a week. Every two weeks, each subject will be admitted to a follow-up visit, during which the physiotherapist will recommend another set of exercises and check the progress. The second group will undergo traditional physiotherapy three times a week for a period of three months. After a period of 3-5 months, both groups will undergo the same examination as initially. The results of both studies will be compared in both groups. The groups will then be compared to each other.

DETAILED DESCRIPTION:
The aim of the study is to compare the effectiveness of individual physiotherapy, using manual therapy, exercises conducted individually and physical therapy to therapy assuming recommendations for self-performed exercises in accordance with the physiotherapist's recommendations. Research questions?

1. Will the effects of self-directed physiotherapy be comparable in terms of reducing pain, improving range of motion, function, and quality of life, and helping reduce the cost of therapy compared to physiotherapy in constant contact?
2. Will the results of subacromial space measurements in ultrasound examination in both groups before and after therapy correlate with clinical and functional tests? The duration of the intervention is assumed at one year. The study will last 3 months. About 60 people will be included in the study, who will be divided into 2 groups, about 30 people each (30 men and 30 women). Patients will be aged 18-50 years. The choice of the group will depend on where the patient comes forward. Patients who report to the Klinika Ruchu will be conducted with individual outpatient physiotherapy - "hands-on". Patients who apply to the Zdrowe Miejsce will be guided by therapy through self-practice "hands off".

The study of patients will include:

1. ultrasound diagnostics,
2. Neer test,
3. palpation of the joint area, taking into account the assessment of the condition of the rotator cuff muscles and muscle around the scapula to exclude possible pronounced atrophy, which may indicate damage to the nerve roots from the C5-6 level, sometimes 7- Erb damage,

3. tests of shoulder mobility according to FMS, 4. cross body abduction stress test to exclude changes in the shoulder-clavicle joint, 5. numerical scale of pain level 0-10, 6. assessment of the pulse on the radial artery in order to exclude damage to the subclavian artery, 7. tension tests of long nerves of the upper kk, 8. DASH Upper Limb Disability Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* age 18-5 0 years,

  * shoulder pain lasting from 3 months to 1 year,
  * no surgery and injection intervention in the shoulder joint and surrounding area in the history of the disease.
  * ailments in scales I and II according to Neer.

Exclusion Criteria:

* surgical procedures and other surgical interventions
* features of the total rupture of the rotator cuff muscle- III⁰ according to Neer scale, confirmed in imaging studies.
* age under 25 or over 50 years
* diagnosed in ultrasound or MRI with complete damage to the muscles of the rotator cuff,
* the duration of the ailment is up to 3 months or more than 1 year.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2023-12-03 (Estimated)

PRIMARY OUTCOMES:
Ultrasound examination | 3 month of observation
  The measurement will be carried out on one ultrasound device. In all patients, a measurement of the subscapular space of the shoulder joint in the ultrasound image will be performed. Ultrasound examinations are used in the diagnosis of the shoulder joint to assess the thickness and quality of tendons and recognized them. Examinations will take place in the positions: of the suspended upper limb and in the position of visit and external rotation in the shoulder joint. Putting on the Power Doppler mesh will allow you to exclude visible inflammation of the examined area while excluding ongoing acute inflammation. In case of doubt or when the examination shows acute inflammation, the patient will be referred to a doctor and a specialist. The measurement will be carried out on one ultrasound device - Siemens Acuson X150, 10-5 MHz linear fisheries. , by one experienced physiotherapist in accordance with the guidelines
Neer test | 3 month of observation
  Performing the test: the subject sits sideways to the examiner, the upper c. of the subject with a bent elbow joint and a bent and brought shoulder joint. The examiner resists the subject's elbow from above, who slightly presses his elbow on the investigator's hand. Results: + pain appears in the test position or after pressure, - no pain, +/- the subject is not able to assess the pain
Palpation. | 3 month of observation
  The examination is carried out in a sitting position with the upper limb suspended.
Shoulder joint mobility according to FMS | 3 month of observation
  The test evaluates the bilateral mobility of the entire shoulder girdle. The test evaluates the bilateral mobility of the entire shoulder girdle, combining internal rotation with arrival and external rotation with visitation. Proper mobility also requires mobility in the shoulder-scapular joint and in the thoracic spine.
Cross-body abduction stress test | 3 month of observation
  The subject sits with a limb bent to 90⁰ in the shoulder and elbow joint. Performs the movement of horizontal attachment in the shoulder joint
The numerical scale of pain level 0-10 | 3 month of observation
  The patient is asked to determine the level of pain on a scale of 0-10. The subject is asked to determine the level of pain on a scale of 0-10, in which it is determined how severe the pain is, indicating the appropriate digit on a scale from 0 to 10, where 0 corresponds - "I do not feel pain at all", - 10 - "the worst pain I can imagine"
Assessment of pulse on the radial artery | 3 month of observation
  Examination is performed to exclude the syndrome stealing of the subclavian artery
DASH Questionnaire | 3 month of observation
  The questionnaire is concerning upper limb disability. The subject assesses his ability to perform the following actions last week by outlining the number of the most accurate answer in Table 1.
  The subject then assesses the severity of symptoms last week by outlining the number in Table 2 of the most accurate answer. After completing the test, we count the sum of points.
  DASH Limitations and Symptoms Index = -1)]×25 where: n = numbers of the answers given. If more than three questions are left unanswered, the DASH cannot be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Kepczynski, Study Director — Klinika Ruchu
Locations (1):
- Klinika Ruchu, Warsaw, Masovian Voivodeship, Poland